CLINICAL TRIAL: NCT03342976
Title: Evaluation of an ICT-based Platform for Early Detection and Intervention to Prevent Frailty in Older Adults
Brief Title: Investigating My Active and Healthy Aging
Acronym: my-AHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Prof. Innocenzo Rainero, Associate Professor of Neurology, University of Turin, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PHC21-2015-689592
Record Dates: First submitted 2017-10-22; First posted 2017-11-17 (Actual); Last update posted 2023-11-30 (Actual); Status verified 2023-11

CONDITIONS: Frail Elderly Syndrome; Cognitive Impairment; Physical Dependence
Keywords: Frailty; Physical impairment; Cognitive decline; ICT
MeSH Terms: conditions — Cognitive Dysfunction; Frailty

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cases (Active Comparator): Pre-frail subjects will use an ICT platform (my-AHA platform) embedded in a mobile phone and a fit-band that will continuously monitor physical and cognitive activities.
  Interventions regarding physical, cognitive, psychological and social domains will be prescribed and monitored through the my-AHA platform. In addition, sleep and dietary habits will be investigated and tailored interventions will be suggested.
  Interventions: Other: My-AHA platform
- Controls (Placebo Comparator): Pre-frail subjects will be followed according to "best standard of care" protocols. Interventions regarding physical, cognitive, psychological and social domains will be prescribed. In addition, sleep and dietary habits will be investigated and tailored interventions will be suggested.
  Interventions: Other: My-AHA platform

INTERVENTIONS:
Other: My-AHA platform — ICT strategy for early detection of frailties

SUMMARY:
This is a multicenter, multicultural, randomized control trial. Participants will be recruited from 10 centers located in Italy, Germany, Austria, Spain, United Kingdom, Belgium, Sweden, Japan, South Korea and Australia. The main objective of the study is to examine the efficacy of a sensor-based platform (my-AHA platform) to assess frailty risks and to deliver tailored interventions in order to prevent in elderly subjects conversion from a pre-frail status to a frailty status.

DETAILED DESCRIPTION:
In the past decade, frailty has attracted great attention of the scientific community and public health organizations as precursor and contributor of age-related diseases. Frailty is a common clinical syndrome in older adults, affecting 7-12% of the older population, and the occurrence of frailty increases with age and may exceed 45% after age 85 years. Frailty develops when age-associated degenerative processes overwhelm reserve capacity and reparative processes that maintain function of the nervous system as well as other physiologic systems. Overall, frailty consists in the vulnerability of aged population to adverse events as the result of the subtle and progressive metabolic and physical changes. Frailty confers a significantly increased risk for poor health outcomes, incident disability, hospitalization, and mortality.

In recent years there has been an emergence of information and communication technology (ICT) -based solutions to support active ageing and tackle frailty, cognitive decline and social isolation of older adults. While these ICT-based solutions are of a certain value regarding diminishing single risks (e.g. fall risk, etc.), there is still a need for a more holistic approach which aims to address all of the individual risk factors together. Also it is necessary to provide tailored interventions based on the outcomes of the risk analysis. This assessment of risk for frailty and provision of individual tailored interventions is the main objective of My-AHA project.

My-AHA solution supports active and healthy ageing by enabling early detection and minimization of risks associated with ageing. In these terms the early risk detection considers three fundamental aspects of the life of older adults: physical activity (by considering vital signs data, gait, quality of sleep and in general, physical activity, and fall risk); cognitive activity (by monitor the cognitive level, e.ge.g. in cognitive games); and, psychosocial activities (e.g. by analyzing the emotions and the quality of speech of the users). On the other hand, My-AHA will develop and implement more efficient and effective ICT-based interventions tailored to the early identified risks. The suggested social activities, as well as cognitive and physical trainings and the diet proposed to the older adults via the new platform will help the users in changing their behaviour and in reacting to the consequences of ageing.

ELIGIBILITY:
INCLUSION CRITERIA for pre-screening

1. Age: over 60 yrs
2. Able to stand and walk unassisted
3. Free of significant cognitive impairment (age-corrected Mini Mental State Examination Test ≥ 24)
4. Free of clinically significant mood disturbance (HADS-Anxiety <15; HADS-depression < 15)
5. Free of any acute or unstable medical conditions
6. Able to understand directions and participate in the protocol
7. Able to sign informed consent

Subjects will be enrolled in the study if they meet one or two of the Fried et al. (2001) criteria for Frailty (Pre-Frailty status).

1. Shrinking, evidenced by weight loss (unintentional) ≥ 4.5 kg unintentional in prior 12 months; or at follow-up assessment ≥ 5% of body weight in prior 12 months.

2, Weakness. Grip strength in lowest 20% at baseline adjusted for gender and BMI.

3. Poor endurance and energy. Self-report of exhaustion as indicated by responses to 2 questions on Center for Epidemiologic Studies Depression (CES-D) scale.

4. Slowness .Time to walk 15ft (4.57m) ≤ slowest 20% adjusted for gender and standing height.

5. Low physical activity level. Lowest quintile (25%) by gender for weighted kcal expenditure per week at baseline.

EXCLUSION CRITERIA

Participant excluded if meets 1 or more of below:

Mobility problems

1. cannot stand and ambulate unassisted
2. painful arthritis, spinal stenosis, amputation, or painful foot lesions that limits balance and mobility,

Concurrent chronic disease independently contributing to frailty

1. suffers from a significant neurodegenerative disorder, e.g.

   1. Alzheimer's disease
   2. Lewy body dementia
   3. Frontotemporal Lobar Degeneration, Fronto-Temporal Dementia
   4. Parkinson's disease
   5. multiple sclerosis
   6. progressive supranuclear palsy
   7. amyotrophic lateral sclerosis
   8. hydrocephalus
   9. Huntington's disease
   10. prion diseases
2. affected by severe peripheral nervous system and/or neuromuscular disorders, e.g.

   1. chronic inflammatory demyelinating polyneuropathy
   2. myasthenia gravis
   3. multiple sclerosis
   4. polymyositis

Concomitant injury or disease known

1. clinical evidence or history of stroke (within 2 yrs) to impact independently cognitive,
2. clinical evidence or history of transient ischemic attack (within 6 months) psychological or physical function
3. significant head injury with associated loss of consciousness, skull fracture or persisting cognitive impairment (2 years)
4. epilepsy (a single prior seizure is considered acceptable)
5. if meet Diagnostic and Statistical Manual 5 (DSM-5) criteria for:

   1. major depressive disorder (current)
   2. schizophrenia or other psychotic disorders (lifetime)
   3. bipolar disorder (within the past 5 years
   4. substance (including alcohol) related disorders (within the past 2 years)

Presence of cognitive, sensory or

1. have language deficits that impair testing perceptual deficits that interfere with assessment tasks
2. have significant visual impairment
3. have a significant hearing loss

Presence of other conditions or diseases that will compromise ability to undertake interventions (especially physical)

1. have clinically significant cardiovascular disease, i.e:

   1. hospitalization for acute coronary syndrome (acute myocardial infarction or unstable, angina)
   2. symptoms consistent with angina pectoris, within the 12 months
   3. signs or symptoms of clinical heart failure within the 12 months
   4. evidence of uncontrolled atrial fibrillation
   5. a cardiac pacemaker
2. preexisting or current signs or symptoms of respiratory failure, e.g.

   1. chronic obstructive pulmonary disease
   2. bronchial asthma
   3. lung fibrosis
   4. other respiratory disease
3. untreated hypertension
4. metastatic cancer or immunosuppressive therapy
5. concurrent acute or chronic clinically significant immunologic, hepatic (such as presence of encephalopathy or ascites), or endocrine disease (not adequately treated).

Unacceptable Test/Laboratory Values

1. Postural hypotension (fall in systolic blood pressure of greater than 30 mmHg or fall in diastolic blood pressure of greater than 20 mmHg on standing compared to sitting) at the time of screening. Subjects who present at the time of screening with postural hypotension yet have no known history of postural hypotension, nor underlying medical condition related to hypotension, may be rescreened

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2018-05-03 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Conversion rate from a pre-frail status to a frail status (Fried criteria) | 18 months
  Comparison of conversion rate in cases and controls between pre-frail status fo frail status

CONTACTS AND LOCATIONS:
Overall Officials: Georg Aumayr, PhD, Principal Investigator — Johanniter International; Helios De Rosario, PhD, Principal Investigator — IBV-Gesmed, Spain; Mathew Summers, PhD, Principal Investigator — Sunshine Coast University, Australia
Locations (1):
- Aging Brain and Memory Clinic, Department of Neuroscience, University of Torino, Torino, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Choi J, Ahn A, Kim S, Won CW. Global Prevalence of Physical Frailty by Fried's Criteria in Community-Dwelling Elderly With National Population-Based Surveys. J Am Med Dir Assoc. 2015 Jul 1;16(7):548-50. doi: 10.1016/j.jamda.2015.02.004. Epub 2015 Mar 14. PMID 25783624
- [Background] Kojima G, Taniguchi Y, Iliffe S, Walters K. Frailty as a Predictor of Alzheimer Disease, Vascular Dementia, and All Dementia Among Community-Dwelling Older People: A Systematic Review and Meta-Analysis. J Am Med Dir Assoc. 2016 Oct 1;17(10):881-8. doi: 10.1016/j.jamda.2016.05.013. Epub 2016 Jun 17. PMID 27324809
- [Background] Shamliyan T, Talley KM, Ramakrishnan R, Kane RL. Association of frailty with survival: a systematic literature review. Ageing Res Rev. 2013 Mar;12(2):719-36. doi: 10.1016/j.arr.2012.03.001. Epub 2012 Mar 12. PMID 22426304
- [Background] Panza F, Solfrizzi V, Frisardi V, Maggi S, Sancarlo D, Adante F, D'Onofrio G, Seripa D, Pilotto A. Different models of frailty in predementia and dementia syndromes. J Nutr Health Aging. 2011 Aug;15(8):711-9. doi: 10.1007/s12603-011-0126-1. PMID 21968870
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156

DOCUMENTS (1):
  • Study Protocol (2017-10-22): https://cdn.clinicaltrials.gov/large-docs/76/NCT03342976/Prot_000.pdf